CLINICAL TRIAL: NCT02040389
Title: Visual Guidelines and Tutoring in Pediatric Urological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92/13
Record Dates: First submitted 2014-01-08; First posted 2014-01-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2013-11

CONDITIONS: Hypospadias; Undescended Testis; Hydrocele; Ureteropelvic Junction Stenosis; Anxiety
Keywords: children; penile; inguinal; kidney parents; anxiety
MeSH Terms: conditions — Hypospadias; Cryptorchidism; Testicular Hydrocele; Multicystic renal dysplasia, bilateral; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pictures book + standard education (Active Comparator): arm with children undergoing urological procedures and their parents will receive standard preoperative education + pictures book with pictures of surgical wound in different stages of healing
  Interventions: Behavioral: Picture book
- Standard preoperative education (Active Comparator): Arm with children undergoing urological procedures and their parents will receive only standard preoperative education
  Interventions: Behavioral: Standard preoperative education

INTERVENTIONS:
Behavioral: Picture book — Arm with showing and explaining for parents about perioperative typical surgery site/wound view by study's team
  Arms: pictures book + standard education
Behavioral: Standard preoperative education — Arm with standard, verbal explaining for a parents about perioperative site/wound view
  Arms: Standard preoperative education

SUMMARY:
The aim of this study is checking impact of visual guidelines (picture book) and tutoring in pediatric urologic surgery

DETAILED DESCRIPTION:
The number of operations in pediatric urology performed on the basis of one day surgery has been increased tremendously over the last years. The shortening of the hospital admission intends to increase the efficacy of the health system, however at the same time puts an additional burdening regarding the postoperative care on the parents of the operated children. The parents often have no or has little experience with regards to the basic medical education. The lack of the proper tutoring in terms of possible complications, normal postoperative period may cause unnecessary patients and parents anxiety, visit to the emergency room or calls to the medical stuff, and in some case delay medical attention which can cause major surgery related complications. Visual guidelines and tutoring of the patients upon surgery may avoid these undesirable effects of the early hospital discharge

Patients and methods:

The investigators are proposing prospective study of 3 groups of patients which undergo the most often urological surgery Group 1 penile surgery, Group 2 inguinal surgery. Group 3 renal surgery required nephrostomy tube leave or drainage. Each group will be divided into two subgroups (20 patients each) with and without visual tutoring prior to the surgery. Visual tutoring will include the photograph pictures reflecting different stage of the convalescent period following surgery. The parents will be asked to answer on questionnaire regarding the level of anxiety before surgery, immediately after surgery, week and 3-6 months after surgery. The number of parents calls to the hospital staff, emergency or outpatient clinic visit will be recorded and compared between two groups. The statistical analysis will performed utilizing Graph Pad Prism version 5.00 for Windows, (Graph Pad software, San Diego, California, chi square and Fisher test), considering p value of <0.05 as significant).

ELIGIBILITY:
Inclusion Criteria:

* children with indications for penile, inguinal or kidney surgery

Exclusion Criteria:

* prior urological procedure (recurrent cases)

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Level of parents anxiety | Thirty minutes before surgery
  The following parameters will be compared between two groups: level of parents anxiety by questionnaire, numbers of parents calls to the hospital staff and non-planed visits to emergency department/outpatient clinic
Level of parents anxiety | Fifteen minutes after surgery
  Measuring of parents anxiety in recovery room after surgery
Level of parents anxiety | Week after surgery
  Measuring of parents anxiety one week after surgery
Level of parents anxiety | Three weeks after surgery
  Measuring of parents anxiety 3-6 weeks after surgery

SECONDARY OUTCOMES:
Numbers of parents non-planed calls/visits | During a week before surgery
  We will note in two groups all non-planned calls/visits before surgery
Numbers of parents non-planed calls/visits | During 48 hours after surgery
  We will note in two groups all non-planned calls/visits during 48 hours after surgery
Numbers of parents non-planed calls/visits | 0ne week after surgery
  We will note in two groups all non-planned calls/visits one week after surgery
Numbers of parents non-planed calls/visits | During 3-6 weeks after surgery
  We will note in two groups of patients all non-planed calls/visits 3-6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Boris Chertin, MD, Prof., Study Chair — Head, The Department of Pediatric Urology, Shaare Zedek Medical Center, Clinical Professor in Surgery/Urology, Faculty of Medicine, Hebrew University, Jerusalem, Israel
Locations (1):
- The Department of Pediatric Urology, Shaare Zedek Medical Center, Faculty of Medicine, Hebrew University, Jerusalem, Israel

REFERENCES:
- [Background] Ono S, Oikawa I, Hirabayashi Y, Manabe Y. Preparation of a picture book to support parents and autonomy in preschool children facing day surgery. Pediatr Nurs. 2008 Jan-Feb;34(1):82-3, 88. No abstract available. PMID 18361093
- [Background] Nelson CP, Rosoklija I, Grant R, Retik AB. Development and implementation of a photographic atlas for parental instruction and guidance after outpatient penile surgery. J Pediatr Urol. 2012 Oct;8(5):521-6. doi: 10.1016/j.jpurol.2011.09.012. Epub 2011 Oct 20. PMID 22018934
- [Background] Moix J, Bassets J, Caelles RM. [Effectiveness of audiovisual materials as a preparation for surgery in pediatric patients]. Cir Pediatr. 1998 Jan;11(1):25-9. Spanish. PMID 9662867